CLINICAL TRIAL: NCT05340673
Title: A Randomized Clinical Trial Comparing Supplemental Topical Treatments for Acute Radiation Dermatitis in Breast Cancer Patients
Brief Title: Comparing Supplemental Topical Agents for the Treatment of Acute Radiation Dermatitis in Patients With Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21152; NCI-2022-01957 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21152 (Other: City of Hope Medical Center); P30CA043703 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Aquaphor) (Experimental): Beginning on day 1 of radiation therapy, patients apply Aquaphor BID, but not within the four hours before EBRT, to the irradiated field until 2 weeks following completion of EBRT.
  Interventions: Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Miaderm) (Experimental): Beginning on day 1 of radiation therapy, patients apply Miaderm BID, but not within the four hours before EBRT, to the irradiated field until 2 weeks following completion of EBRT.
  Interventions: Drug: Agent Affecting Integumentary System; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Agent Affecting Integumentary System — Apply Miaderm
  Arms: Arm II (Miaderm)
Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment — Apply to skin
  Other Names: Aquaphor
  Arms: Arm I (Aquaphor)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares two supplemental topical agents (Aquaphor and Miaderm) for the treatment of acute radiation dermatitis in patients with breast cancer undergoing radiation therapy. Radiation dermatitis is a radiation-induced skin reaction which can cause itching, swelling, pain, and general discomfort. Aquaphor is a commonly available, inexpensive, petrolatum-based multi-purpose ointment designed to protect and sooth extremely dry skin, chapped lips, cracked hands and feet, minor cuts and burns, and many other skin irritations. Miaderm is a water-based cream and contains ingredients like calendula, hyaluronate, and aloe vera which may help reduce occurrence and severity of radiation dermatitis. Both are commonly recommended and used by breast cancer patients undergoing external beam radiation therapy (EBRT). However, it is not known whether one is better than the other in treating or preventing radiation dermatitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of Miaderm compared to Aquaphor in the treatment and/or prevention of radiation dermatitis caused by EBRT in breast cancer patients undergoing EBRT to the breast/chest wall.

SECONDARY OBJECTIVE:

I. Determine quality of life (QoL) and need for additional concomitant therapies to address dermatitis in breast cancer patients undergoing EBRT to the breast/chest wall using Miaderm compared to Aquaphor.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning on day 1 of radiation therapy, patients apply Aquaphor twice daily (BID), but not within the four hours before EBRT, to the irradiated field until 2 weeks following completion of EBRT.

ARM II: Beginning on day 1 of radiation therapy, patients apply Miaderm BID, but not within the four hours before EBRT, to the irradiated field until 2 weeks following completion of EBRT.

After completion of study treatment, patients are followed up at 2 weeks and then at 90-120 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.
* Age > 18 years.
* Undergoing external beam radiation therapy (EBRT) to the breast or chest wall following surgical resection (lumpectomy or mastectomy) for ductal carcinoma in situ (DCIS) or invasive breast cancer using either conventional fractionation or hypofractionation.

Exclusion Criteria:

* Partial breast irradiation.
* Prior radiation overlapping with the intended radiotherapy field.
* History of systemic radiation sensitivity diseases (xeroderma pigmentosum, ataxia telangiectasia).
* Extreme hypofractionation (less than 15 fractions of radiation).
* Palliative treatment.
* Patient intention to use topical product other than Aquaphor or Miaderm.
* Inflammatory breast cancer, skin involvement, planned use of bolus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Acute Radiation Dermatitis | Up to 120 days after completion of radiation therapy
  Depending on prescribed duration of radiation treatment, each subject will contribute between 5 and 8 periodic assessments for the presence of acute radiation dermatitis Radiation Therapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG/EORTC toxicity score of 2 or higher). The hypothesized association between randomized treatment and the repeated binary outcome of Acute Radiation Dermatitis will be tested using repeated measures logistic regression. That model will be implemented with PROC GENMOD (SAS software) for a generalized linear regression model with generalized estimating equation (GEE) for binary data with logit link function. In this way, the analysis will recognize the within-patient correlation inherent in repeated assessments.

SECONDARY OUTCOMES:
Quality of life (QoL) | Up to 120 days after completion of radiation therapy
  Skindex-16 is a single-page, validated measure of the effects of skin disease on patients' quality of life. The 16 questions address Symptoms (4 items), Emotions (7 items), and Functioning (5 items). Using a 7-level scale that is scored from 0 (Never bothered) to 100 (Always bothered), each question asks how much during the last 7 days the patient has been bothered by a specific aspect of their disease. Responses are averaged to generate a Global score and 3 domain-specific sub-scores, all ranging from 0 to 100, with higher scores indicating worse disease-related quality of life. Evaluated by the Skindex-16 questionnaire will be compared between the two study arms. T tests will be applied to assess mean differences between arms at each time point.
Supportive measures | Up to 120 days after completion of radiation therapy
  Depending on prescribed duration of radiation treatment, each subject will contribute between 5 and 8 periodic assessments for the use of Concomitant Therapy for acute radiation dermatitis. The hypothesized association between randomized treatment and the repeated binary outcome of Concomitant Therapy will be tested using repeated measures logistic regression. Similar to the analysis of the Primary Endpoint described above, this model will be implemented with PROC GENMOD (SAS software) for a generalized linear regression model with GEE for binary data with logit link function and will consider potential covariates and possible treatment-by-time interaction as described above for the Primary Endpoint analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Glaser, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States